CLINICAL TRIAL: NCT05723978
Title: Selective Extended Dissection in Different Types of Pancreatic Head Cancer: A Retrospective Cohort Study.
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Panc-2023129
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Selective extended dissection (SED) group
  Interventions: Procedure: Selective extended dissection of pancreaticoduodenectomy
- Standard dissection (SD) group

INTERVENTIONS:
Procedure: Selective extended dissection of pancreaticoduodenectomy — An optimized procedure of pancreaticoduodenectomy which is based on the extra-pancreatic nerve plexus (PLX) potentially invaded by tumor.
  Groups: Selective extended dissection (SED) group

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is a highly malignant tumor with relatively poor survival. Surgery is the first choice for the treatment of patients with early pancreatic cancer. However, the surgical approach and the extent of resection for patients with pancreatic cancer are controversial at present.

The investigators optimized the procedure of standard pancreaticoduodenectomy to selective extended dissection (SED), which is based on the extra-pancreatic nerve plexus (PLX) potentially invaded by tumor. The investigators retrospectively analyzed the clinicopathological data of patients with pancreatic adenocarcinoma who underwent radical surgery in our center from 2011 to 2020. Patients who underwent standard dissection (SD) were matched 2:1 to those who underwent SED using propensity score matching (PSM). The log-rank test and cox regression model were used to analyze survival data. In addition, statistical analyses were performed for the perioperative complications, postoperative pathology and recurrence pattern.

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients diagnosed as resectable pancreatic cancer were pathologically diagnosed as PDAC after surgery.

2) Patients received radical surgery (R0) and had complete photos or videos of the operation.

Exclusion Criteria:

- 1) The operation records as well as related photo or video data could not reflect the surgical approach and the extent of resection.

2) Patients with incomplete clinical, pathological, imaging and follow-up information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed as resectable pancreatic cancer were pathologically diagnosed as PDAC after surgery
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From the day the patient received surgery to the time the patient was diagnosed with postoperative recurrence, assessed up to 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Guo X, Song Y, Xu P, Zhu W, Wang H, Zhou Y, Huang C, Hao J, Gao S. Selective extended dissection for pancreaticoduodenectomy is associated with better survival in pancreatic cancer patients: retrospective cohort study. Int J Surg. 2023 Jul 1;109(7):1852-1862. doi: 10.1097/JS9.0000000000000437. PMID 37195787